CLINICAL TRIAL: NCT07142447
Title: Understanding and Preventing the Impact of Endocrine Disruptors on the Hypothalamus-pituitary Axis in Sensitive Populations. Hypiend- Perinatal Study.
Brief Title: Effectiveness of a multicOmpoNent Behavioural intervenTion to Reduce endocrINe disrUptor Exposure During pErinatal Period (CONTINUE)
Acronym: CONTINUE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut Germans Trias i Pujol (Other)
Collaborators: KU Leuven (Other); Universidad de Granada (Other); Fundació Eurecat (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 101137440
Record Dates: First submitted 2025-07-24; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Pregnancy; Children
Keywords: Endocrine Disruptors; hormones
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: HYPIEND aims at evaluating whether a multi-centric, multicomponent interventional trial (digital tool aimed at promoting lifestyle habits to reduce EDC exposure by providing personalized recommendations + phone calls + workshops about environmental health education) carried out in 810 women from pregnancy until their children are 18 months old is able to reduce the exposure to different EDCs.
  This intervention will be designed considering the gradual introduction of small changes (i.e., by using goal setting), carrying out a family-based approach, in a personalized manner, considering targeting different routes of exposure and providing to the participants frequent feedback and support. With this design, we expect to promote a behavioural change to achieve long-lasting effects in reducing the exposure to EDCs. The effects will be compared with a control intervention group, which will only receive a digital printable booklet with information on EDC hazards.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral intervention (Experimental): Healthy pregnant women who will receive a multi-component behavioral intervention (digital tool aimed at promoting lifestyle habits to reduce EDC exposure by providing personalized recommendations + telephone monitoring + workshops about environmental health education) during pregnancy and the first 18 months after delivery.
  Interventions: Behavioral: Multi-Component Behavioral intervention
- Control group (Other): Healthy pregnant women who will receive the standard of care. The control condition consists of a single online education module/written information about EDCs addressed to reduce their exposure. They will also have access to the digital tool to answer the questionnaires, but this group will not receive any recommendations or missions from the professionals concerning EDCs along the study. After finishing the intervention, the participants of the control group will be offered access to all the developed material (workshops…) and to use the app.
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Multi-Component Behavioral intervention — A multicomponent behavioral intervention during pregnancy and up to the first 18 months after delivery, composed by:
  1. Digital tool called "App Hypiend Digital Tool" aimed at promoting lifestyle habits to reduce EDC exposure by providing personalized recommendations
  2. Telephone monitoring
  3. Workshop about environmental health education
  Arms: Behavioral intervention
Behavioral: Control group — Minimal behavioral intervention. Usual care
  Other Names: Minimal behavioral intervention. Usual care
  Arms: Control group

SUMMARY:
The general objective of HYPIEND is to understand the effects of chemical substances called "endocrine disruptors" (EDCs) during the perinatal and pre-pubertal stages. EDCs co-exposure may affect the function of hormones and determine endocrine consequences in vulnerable populations.

The primary objective of this clinical study is to demonstrate that a multicomponent intervention implemented in health care centres from three European countries is effective in reducing the levels of EDCs in different body fluids of pregnant women, breastfeeding and formula feeding women as well as in their infants up to 18 months of age, improving at the same time the level of HAPA constructs (psychological determinants of behaviour) and the knowledge about these chemicals at family level.

DETAILED DESCRIPTION:
Study rationale

1. Extent and evaluation of current knowledge directly linked to the scientific question(s) to be answered by the clinical study.

   Human epidemiological data suggest that EDC exposure during the perinatal period can negatively affect infant growth trajectory and neurodevelopment and possibly play an important role in the rapid epidemiological growth of obesity and diabetes. As an example, one study carried out in 460 mother-infant pairs from Korea showed that Mental and/or Psychomotor Developmental Indices of the Bayley Scales of Infant Development were inversely correlated in 6-month-old males with the maternal urinary levels of the phthalate metabolites MEHHP, MEOHP and MBP at the third trimester of pregnancy. Very recently, it was reported that mothers with overweight displayed increased levels of the highly persistent environmental chemicals polychlorinated biphenyls in breast milk 2-weeks postpartum and that there was a negative association between some of these compounds and the head circumference-for-age, weight-for-age, and weight-for-length z-scores of the infant at the age of 6 months.

   However, there are discrepancies among findings, which can be attributed to differences in the temporal window of EDC exposure assessment (i.e., early versus late gestation or lactation), in the infants' age at which the measurements were carried out or to a misclassification of EDC exposure due to a single-point analyses of their exposure. In fact, one of the limitations of many epidemiological studies is the use of single spot urine samples at one time-point to estimate the exposure to EDCs. The limitation relies on the short biological half-lives of many of these chemicals and their quick excretion in urine, properties that cause a demand for multiple time point for a precise estimation of exposure assessment. Although different epidemiological studies have found an association between higher exposure to EDCs and neuroendocrine and neurodevelopmental alterations in toddlers and children, as far as we know, no clinical interventions have been carried out to elucidate whether reducing the exposure to EDCs can contribute to counteract/ameliorate these harmful effects.

   So far, very few human intervention studies focused on reducing the exposure to EDCs during the perinatal period have been conducted, some carrying out educational approaches and others focused on dietary or other changes. Relevantly, most of them had small sample sizes (<100 people) and analysed a maximum of two different types of EDCs and quite a few were carried out without control groups. Moreover, the level of adherence in this type of interventions is low in general, reflecting the need to implement adequately behavioural change techniques to foster long-term lifestyle habit improvements.
2. Outcomes (efficacy, safety) Of completed and number of ongoing clinical studies utilizing the same intervention in the same indication (including review of public registers)

   Recently, the PREVED project was carried out to improve knowledge, to enhance risk perception and to change exposure behaviour regarding EDCs of 268 women during pregnancy and up to 14 months after birth . The authors reported a significant increase in the evolution of risk perception score and overall psychosocial score in the two intervention groups that received 3 workshops during pregnancy, one group in neutral location (leaflet on EDCs and collective workshops in a meeting room), and the other group in contextualized location (leaflet on EDCs and collective workshops in the real-life pedagogical apartment) when compared with a control group (leaflet on EDCs). However, no differences in consumption of canned food and in percentage of women having a decrease in bisphenol A or parabens concentrations in urine were found between the control and the two intervention groups. In another RCT carried out in 51 women in Korea, a 4-week web-based behavioural intervention reduced the urinary concentrations of BPA, different phthalate metabolites, and parabens in mothers with young children . Moreover, an ongoing study aims to determine if a personalized mobile intervention is able to reduce the exposure to EDCs in adults of child-bearing age (ClinicalTrials ID: NCT05780047). Despite some promising results, these examples illustrate the need to carry out larger multicomponent clinical and community-based intervention studies focused on minimize the exposure to EDCs at short, medium, and long time to obtain results that are more conclusive.
3. Level of evidence related to the mechanism of action of the intervention in the planned clinical study population

EDC-Mix-Risk and ENDpoiNTs are two outstanding Horizon 2020 projects that combined the experimental research in both cells and animals with epidemiological data. Researchers of both projects and others nicely showed using a statistical model for multivariate regression with data obtained in the SELMA pregnancy study that different EDCs (including phthalates, alkyl phenols, and perfluoroalkyl substances) analysed in the urine and serum of women at week 10 of pregnancy were associated with language delay of their children at 2.5 years of age. Afterwards, the identified EDCs were mixed and tested in human brain organoids as well as in Xenopus leavis and Danio rerio to elucidate the molecular and functional impact of exposure. Finally, the authors integrated both experimental and epidemiological data and carried out a risk assessment approach, finding increased odds of language delay in up to 54% of the offspring who had prenatal exposures above experimentally derived levels of concern: Despite these very relevant findings, a limited number of studies carried out in humans have shed light on the mechanisms underlying the EDC-mediated dysfunctions on HP axis, including the induction of epigenetic changes in key genes involved in foetal development, neuroendocrine regulation and early puberty as well as the alterations of the inflammatory response and the gut microbiota (dysbiosis). EDCs may increase the risk of childhood neurodevelopmental disorders by interfering with early life estrogenic and thyroid hormone signalling or metabolism. In this sense, in humans, it has been shown that some phthalates may reduce thyroxine and triiodothyronine concentration in pregnant women and children and that the exposure to phthalates produced oxidative stress and can also affect the health of the offspring through epigenetic re-programming of the foetus and placenta. In another study, maternal exposure to heavy metals affected progeny neurodevelopment, and changes in DNA methylation of genes controlling neurodevelopment were observed in cord blood, but not the blood collected at mid-childhood. Analysis of exposure-outcome identified differentially methylated CpG on DAB Adaptor Protein 1 (DAB1) gene as a marker of the effect of prenatal polycyclic aromatic hydrocarbon (PAH) exposure on children's mental development. Increased exposure to PAHs during pregnancy was positively correlated with the methylation of insulin-like growth factor IGF1 and 2, key factors in human growth and development that are maternally imprinted. Incorrect methylation of those genes during early development relates to reduced birth weight and increased predisposition to metabolic problems, like obesity, cardiovascular diseases or diabetes. However, despite this evidence, as far as we know, no human intervention studies aimed at reducing the exposure to EDCs have analysed the molecular impact that can accompany these changes in EDC exposure. Further research is needed to shed more light on these issues, including molecular and omics-based analyses in humans to elucidate whether human intervention studies aimed at reducing EDC exposure can favourably modulate these molecular changes.

Different molecular and omics approaches will be carried out to shed more light in the framework of the HP axis on the epigenetic drivers most susceptible to disruption, the genes and the pathways most differently affected, the interplay between intestinal microbiota and the impact of EDC exposure on systemic inflammation. These analyses will be carried out in samples obtained in the study considering our results obtained in preclinical models exposed to EDC mixtures trying to resemble the real human exposure, to increase the chance to obtain robust and reliable results using a targeted approach. Specifically, in women the analyses will be carried out during pregnancy and after delivery at different time points and will be focused on the analyses of HP axis-related hormones and cytokines, intestinal microbiota, methylation of different CpG sites of key genes involved in HP axis as well as the expression of these genes. In their offspring, in addition to these analyses, the circulating levels of kisspeptin will be also analysed at birth (cord blood) and at the age of 18 months (capillary blood/dry blood spots -DBS-). Overall, these analyses will allow us to go into depth on the mechanisms by which EDCs exert their harmful effects as well as how intervention studies aimed at reducing the exposure to these chemicals can modulate these biological pathways and the molecular biomarkers of exposure identified. As far as we know, this approach has not yet been carried out in large human intervention studies in the framework of EDCs.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with a viable pregnancy confirmed by ultrasound until 13 weeks and 0 days of gestation (recruitment between 6-11 weeks). Their partners will be invited to participate but this is not mandatory for inclusion.
* BMI at Visit 1 between 18.5-40 kg/m²
* Intention to breastfeed
* Being able to read the language of their respective countries (Dutch/French -Belgium-, Spanish and/or Catalan -Spain- and Polish -Poland)
* Being 18 years or older
* In possession of a smartphone. If participants do not have a smartphone because of socio-economic reasons, a smartphone will be at their disposal for the whole duration of the study

Exclusion Criteria:

* Unable to sign informed consent (cultural barriers, psychological conditions)
* Abuse of substances (alcohol, drugs)
* Chronic use (at least, for three months before pregnancy) of any medication that might affect the HP axis:
* Antidepressants
* Insuline.
* Levothyroxine, Methimazole, Propylthiouracil.
* Oral corticosteroids (topical and inhalation formulations will be allowed)
* Arginine vasopressin (AVP)
* Mifepristone.
* Anticortisolic drugs: Metyrapone (Metopirone), Ketokonazole, Osilodrostat (Isturisa), Mitotane (Lysodren), aminoglutethimide (Cytadren) and Levoketoconazole (Recorlev).
* Multiple gestation
* Type 1 or 2 diabetes
* Pregnant women will not be consented into research by any HCP with whom they have a dependent relationship (Declaration of Helsinki) (I would remove this point).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 810 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Decrease of mono(2-ethyl-5-oxohexyl) phthalate (MEOHP) concentration in urine | From first trimester of pregnancy to 18 months after delivery
  This election was based on a scientific article in which was reported that mental and/or Psychomotor Developmental Indices of the Bayley Scales of Infant Development were inversely correlated in 6-month-old infants with the maternal urinary levels of MEHHP and MEOHP at the third trimester of pregnancy in a study carried out with 460 mother-infant pairs (4). However, since during the initial phase of the project a predictive modelling approach will be carried out in order to select the EDC mixtures with high harmful effects to be evaluated in preclinical models, the definitive main outcome could be redefined once we obtain the predictive modelling results.
  We would expect to detect a 25% decrease in the urinary levels of MEOHP in the intervention group vs control group at the end of the study.

OTHER OUTCOMES:
Reduction of EDC levels in biological fluids | From first trimester of pregnancy to 18 months after delivery
  Other EDCs in urine, peripheral blood, cord blood and milk

CONTACTS AND LOCATIONS:
Overall Officials: Inés Velasco, MD, PhD, Principal Investigator — Foundation Institute of Research in Health Sciences Germans Trias i Pujol
Locations (1):
- Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
All data will be treated confidentially, and privacy of all participants will be protected by saving personal data separately from research data on encrypted files with identification numbers that can only be accessed by the main researchers working on this project. The file containing personal data will be destroyed after data collection has been completed. Data about the usage of the application will not contain IP address information and therefore it cannot directly identify its user and related personal information. Data management and agreements to transfer data/samples is dealt in a Data Protection Impact Assessment.

REFERENCES:
- [Background] Schulz MC, Sargis RM. Inappropriately sweet: Environmental endocrine-disrupting chemicals and the diabetes pandemic. Adv Pharmacol. 2021;92:419-456. doi: 10.1016/bs.apha.2021.04.002. Epub 2021 Jun 9. PMID 34452693
- [Background] Heindel JJ, Howard S, Agay-Shay K, Arrebola JP, Audouze K, Babin PJ, Barouki R, Bansal A, Blanc E, Cave MC, Chatterjee S, Chevalier N, Choudhury M, Collier D, Connolly L, Coumoul X, Garruti G, Gilbertson M, Hoepner LA, Holloway AC, Howell G 3rd, Kassotis CD, Kay MK, Kim MJ, Lagadic-Gossmann D, Langouet S, Legrand A, Li Z, Le Mentec H, Lind L, Monica Lind P, Lustig RH, Martin-Chouly C, Munic Kos V, Podechard N, Roepke TA, Sargis RM, Starling A, Tomlinson CR, Touma C, Vondracek J, Vom Saal F, Blumberg B. Obesity II: Establishing causal links between chemical exposures and obesity. Biochem Pharmacol. 2022 May;199:115015. doi: 10.1016/j.bcp.2022.115015. Epub 2022 Apr 5. PMID 35395240
- [Background] O'Shaughnessy KL, Fischer F, Zenclussen AC. Perinatal exposure to endocrine disrupting chemicals and neurodevelopment: How articles of daily use influence the development of our children. Best Pract Res Clin Endocrinol Metab. 2021 Sep;35(5):101568. doi: 10.1016/j.beem.2021.101568. Epub 2021 Sep 4. PMID 34565681
- See also: Official website of the interventional study — https://hypiend.eu/

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-08-21): https://cdn.clinicaltrials.gov/large-docs/47/NCT07142447/Prot_SAP_ICF_000.pdf